CLINICAL TRIAL: NCT00188292
Title: Screening for HIV-Associated Anal Cancer
Acronym: TRACE
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Collaborators: Ontario HIV Treatment Network (Network); Canadian Foundation for AIDS Research (CANFAR) (Other)
Responsible Party: Sponsor
Other Study IDs: REB #02-0325-B; #016005 (Other Grant/Funding Number: CANFAR)
Record Dates: First submitted 2005-09-09; First posted 2005-09-16 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-03

CONDITIONS: HIV Infections; Anal Cancer; Anal Dysplasia; Papillomavirus Infections
Keywords: Human Papillomavirus; Anal; Cancer screening; Immunodeficiency; HIV
MeSH Terms: conditions — HIV Infections; Anus Neoplasms; Papillomavirus Infections; Immunologic Deficiency Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- High-grade disease: Those who had histologic anal high-grade disease.
- Control: Those who had less than highgrade histologic anal disease

SUMMARY:
Cancer of the anus occurs at very high rates in young men with HIV and is caused by a virus called human papillomavirus (HPV). Anal cancer has increased during the HIV epidemic despite effective therapies for HIV. Unfortunately, anal cancer presents at a late stage because there is no screening program to find it at an early stage.

Rates of other cancers such as cervical cancer have been reduced through the use of Pap smears. The researchers' plan is to do the same type of screening for anal cancer as has been done for cervical cancer. If abnormalities are found then treatment can be started. The researchers hope that this approach will help to prevent anal cancer.

Testing for HPV will also be done to see if this helps to detect early cancer and to see how accurate different tests, pathologists and clinical examiners are at detecting and agreeing on any abnormalities.

The main outcome is the presence of any pre-cancerous or early cancer changes as determined by high resolution anoscopy (HRA). HRA involves looking through a microscope into the anus and this allows very tiny changes to be identified. Pieces of tissue can then be taken to make a definite diagnosis.

DETAILED DESCRIPTION:
Anal cancer occurs at a rate which is 163-fold greater in young men with HIV. It is caused by another virus, HPV. The incidence has doubled during the HIV epidemic and is not decreasing despite effective antiretroviral therapy. It is important to have an anal cancer screening program to detect precancerous lesions; this has been done for the prevention of cervical cancer through the use of cervical Pap smears.We will do anal Pap smears, HPV testing and perform high resolution anoscopy for a magnified and detailed view of the anus. Biopsies are done and early treatment is initiated. It is anticipated that this approach will help to prevent anal cancer.

SPECIFIC AIMS:

The aim of this study is to determine the accuracy of pathology and human papillomavirus (HPV) testing in identifying precancerous changes in HIV positive men. The primary question is to determine how good the anal Pap smears are for detecting precancerous changes in the anus. Secondary questions involve: (a) determination of the test characteristics of the anal Pap smear, (b) assessment of agreement in visually detecting pre-cancers by the anoscopists and, (c) a determination of the viral and patient characteristics that predict pre-cancer.

STUDY DESIGN:

This is a cross-sectional survey of HIV positive men with a history of anal receptive intercourse who are attending several Toronto HIV clinics. Relevant information is collected as well as anal specimens for assessment. There is a multidisciplinary team who have the appropriate expertise in these studies.

OUTCOME MEASURES and STATISTICAL ANALYSIS:

The primary outcome measure is the presence of pre-cancerous changes as determined by high resolution anoscopy. We need to screen 425 subjects in order to find 100 patients with high grade pre-cancerous changes.

Secondary outcome analyses include specificity, positive predictive value and negative predictive value of cytology and HPV DNA testing to detect histologically confirmed pre-cancerous changes or cancer.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected men,
* History of anal receptive intercourse,
* Minimum age 18 years.

Exclusion Criteria:

* Known anal cancer,
* Bleeding diathesis that might preclude anoscopy and biopsy.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV + MSM who had High Resolution Anoscopy
Sampling Method: Probability Sample
Enrollment: 401 (Actual)
Dates: Start 2002-08; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Irving E Salit, MD, Principal Investigator — Toronto General Hospital
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada